CLINICAL TRIAL: NCT04388358
Title: Study the Effects of Traditional Chinese Medicine for the Treatment of Perennial Allergic Rhinitis on Gut Microbiota and Immune-modulation in Humans
Brief Title: Traditional Chinese Medicine for the Treatment of Perennial Allergic Rhinitis on Gut Microbiota and Immune-modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, YANG SIEN-HUNG, Director of Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMRPD1J0771
Record Dates: First submitted 2020-05-07; First posted 2020-05-14 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Allergic Rhinitis
Keywords: Perennial allergic rhinitis; Gut microbiota; Mixe formula of Chinese medicine
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Perennial | interventions — sho-seiryu-to

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mixed Chinese herb formula (Other): Shin-yi-san + Xiao-qing-long-tang + Xiang-sha-liu-jun-zi-tang by the weight of 9g+3g+3g/day
  Interventions: Drug: Shin-yi-san + Xiao-qing-long-tang + Xiang-sha-liu-jun-zi-tang by the weight of 9g+3g+3g/day

INTERVENTIONS:
Drug: Shin-yi-san + Xiao-qing-long-tang + Xiang-sha-liu-jun-zi-tang by the weight of 9g+3g+3g/day — All patients were treated with mixed formula of Chinese medicine for one month

SUMMARY:
40 allergic rhinitis patients in the acute phase will be enrolled in the study. All the allergic patients should be confirmed those who are over 20 years old and hypersensitive to house dust mite allergens confirmed by MAST test before study. All patients were treated with mixed formula of Chinese medicine for one months.

DETAILED DESCRIPTION:
Perennial allergic rhinitis is an important disease in traditional Chinese medicine (TCM) due to its high prevalence rate in Taiwan. In our previous studies, a new mixed formula of Chinese herbs was evaluated for the treatment of allergic rhinitis. In these studies, we found that immunoduoatory effects of Chinese medicine include: CD4+ T lymphocytes; Regulatory T cells; Dendritic cells, and Regulatory B cells. These results allow us to confirm the immunomodulatory effects of mixed formula of traditional Chinese medicine. In recent years, more and more attention has been paid to the effects of gut microbiota on immune-modulation. Many immunomodulaotry effects of allergic diseases were considered to be closely related to gut bacteria. However, the research on allergic rhinitis is still rare, especially related to TCM treatment. From our previous studies, it has been confirmed that TCM have an immunomodulatory effect on allergic rhinitis. Whether or not they are associated with gut microbiota changes is still unknown. This year, we compared the difference of composition and diversity of gut microbiota of allergic rhinitis patients and normal individual. Indeed, we found it were different between allergic patients and normal individuals. The results of this study will provide us the information to understand whether the immunemodulation of TCM treatment on allergic rhinitis is correlated with the changes of gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer for study enrollment and sign inform consent
* Mite allergy confirmed by MAST test
* Over 20 years old
* Will have their blood collected twice and stool samples
* Allergic rhinitis patients in the acute phase will be treated with mixed formula of Chinese medicine for one months

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Under treatment of western medicine including steroid, antihistamine, leukotriene inhibitor, immunosuppressant or stop above medication less than one month
* Under acute inflammatory disease such as pneumonia, sinusitis, bronchitis and so on vasomotor type allergic rhinitis
* History of allergy or adverse effect to Chinese herbs, poor compliance of herbal medicine severe organ function impairment, such as heart failure, liver failure, renal failure (eGFR <60 mL/min/1.73 m2)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Serum IgE level assessments and MAST test | On starting day (day 0)
  check serum total IgE and mite specific IgE

SECONDARY OUTCOMES:
CD4+ Cell isolation and purification | Assessment of CD4+ on Day 0 and 1 month after completing treatment
  check CD4 Cell by flowcytometry
Quantification of mRNA expression by means of RT-PCR and real-time PCR | Assessment of mRNA on Day 0 and 1 month after completing treatment
Gut microbiota data analysis procedures | Assessment of gut microbiota on Day 0 and 1 month after completing treatment
  use cecal stool DNA purification and quantification of cecal microbiota by quantitative PCR (qPCR). Using V3-V5 16S rRNA amplification; Processing of NGS data; Operational Taxonomic Units (OTUs) cluster; Taxonomic profiling

CONTACTS AND LOCATIONS:
Overall Officials: Sien-hung Yang, Ph.D, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided